CLINICAL TRIAL: NCT02416869
Title: Effectiveness of Different Application Modalities of Dexamethasone on Clinical Parameters and Quality of Life After Lower Third Molar Surgery
Brief Title: Dexamethasone in Lower Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Miroslav Andric, Assistant Professor, University of Belgrade
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 36/11-2013
Record Dates: First submitted 2015-04-02; First posted 2015-04-15 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Impacted Third Molar Tooth
Keywords: Dexamethasone; Lower third molar surgery
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Intramuscular application (Active Comparator): Intramuscular application of 4mg Dexamethasone
  Interventions: Procedure: Intramuscular application
- Submucosal application (Experimental): Submucosal application of 4mg Dexamethasone
  Interventions: Procedure: Submucosal application
- 4mg Dexamethasone submucosal (Active Comparator): 4mg Dexamethasone submucosal application
  Interventions: Drug: 4mg Dexamethasone submucosal
- 8mg Dexamethasone submucosal (Experimental): 8mg Dexamethasone submucosal application
  Interventions: Drug: 8mg Dexamethasone submucosal
- 4mg Dexamethasone postoperative (Active Comparator): 4mg Dexamethasone postoperative application
  Interventions: Procedure: 4mg Dexamethasone preoperative
- 4mg Dexamethasone preoperative (Experimental): 4mg Dexamethasone postoperative application
  Interventions: Procedure: 4mg Dexamethasone postoperative

INTERVENTIONS:
Procedure: Intramuscular application — Patient receive 4mg of Dexamethasone by intramuscular application
  Arms: Intramuscular application
Procedure: Submucosal application — Patients receive 4mg of Dexamethasone by submucosal application
  Arms: Submucosal application
Drug: 4mg Dexamethasone submucosal — Patients receive 4mg of submucosal Dexamethasone
  Other Names: Dexasone
  Arms: 4mg Dexamethasone submucosal
Drug: 8mg Dexamethasone submucosal — Patients receive 8mg of submucosal Dexamethasone
  Other Names: Dexasone
  Arms: 8mg Dexamethasone submucosal
Procedure: 4mg Dexamethasone preoperative — Patients receive 4mg of Dexamethasone preoperatively
  Arms: 4mg Dexamethasone postoperative
Procedure: 4mg Dexamethasone postoperative — Patients receive 4mg of Dexamethasone postoperatively
  Arms: 4mg Dexamethasone preoperative

SUMMARY:
The aim of this randomized double-blind cross over clinical trial is to investigate effectiveness of different routes of applications (intramuscular and submucous at the site of surgery) and doses (4 mg and 8 mg) of Dexamethasone on swelling, trismus, pain and quality of life after lower third molar surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (ASA I)
* Bilateral symmetrically impacted lower third molars according to Pel-Gregory's and Winter's classification

Exclusion Criteria:

* Heavy tobacco smokers
* Drug and / or alcohol abusers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Facial swelling (using 3 facial measurements (in millimeters) | 1 day, 3 day, 7 day
  We followed facial swelling 1, 3 and 7 days after intervention.
  Swelling in the operation site will be evaluated using 3 facial measurements (in millimeters):
  1. Tragus - Midline.
  2. Tragus - Corner of the mouth
  3. Gonion - Lateral canthus.

SECONDARY OUTCOMES:
Postoperative pain (visual analog scale) | 1 day, 3 day, 7 day
  Postoperative pain will be evaluated using a visual analog scale, 100 mm in length ranging from 0 for " no pain" to 100 for "the worse imaginable pain".
Postoperative trismus (difference in interincisal distance at the maximal mouth opening (in millimeters) before and after surgery) | 1 day, 3 day, 7 day
  Postoperative trismus will be measured as the difference in interincisal distance at the maximal mouth opening (in millimeters) before and after surgery.
Postoperative discomfort (25-items custom made questionnaire) | 4 day, 7 day
  Postoperative discomfort will be evaluated by filling out the 25-items custom made questionnaire that was designed to asses the patient's perception of adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav M Andric, DDS, PhD, Principal Investigator — University of Zagreb
Locations (1):
- School of Dental Medicine, Belgrade, Serbia